CLINICAL TRIAL: NCT02127346
Title: Relationship Between Chronic Periodontitis and Vitamin D and Calcium in Men
Status: Completed | Type: Observational
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Other Study IDs: UDDS-Perio-04-2014
Record Dates: First submitted 2014-04-25; First posted 2014-04-30 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2015-10

CONDITIONS: Chronic Periodontitis
Keywords: Chronic Periodontitis; Vitamin D concentration; Calcium concentration
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Chronic Periodontitis: 1. Male patients
  2. Patients are suffering from chronic periodontitis
  3. Patients do not have any systemic diseases
  4. Subjects should have 20 teeth at least
  5. Age: 30 years or greater
- Healthy Volunteers: 1. Males
  2. Healthy with no systemic diseases or periodontitis
  3. 30 years old at least
  4. 20 teeth are present at least

SUMMARY:
Objective: The objective was to evaluate whether serum vitamin D and calcium concentrations are associated with chronic periodontitis in Syrian men Methods: This study designed as "Matched Case-Control Study".200 males will be enrolled in this study and will be divided into two groups. First group consist of 100 patients suffering from chronic periodontitis and no systemic diseases. Second group consist of 100 healthy volunteers. Serum vitamin D and calcium concentrations will be tested. Periodontal indexes include probing depth (PD), clinical attachment level (CAL), and bleeding on probing (BOP) will be taken. Data will be collected and analyzed.

DETAILED DESCRIPTION:
Periodontal disease including chronic periodontitis results from interaction between pathogens and the host inﬂammatory response. This interaction triggers a complex process of inﬂammatory events, which in turn promote connective tissue destruction and alveolar bone remodeling. Periodontitis is described as a multifactorial irreversible and cumulative condition, initiated and propagated by bacteria and host factors.

Vitamin D and calcium are fundamental for bone mineralization and for the prevention of osteoporosis Severe vitamin D deficiency lead to mineralization defects but chronically low intake of vitamin D and calcium leads to bade calcium balance and bone loss, and it is reasonable to expect this effect to occur in alveolar bone as it does in other bones of the body. A study has showed a positive association between low bone mass or osteoporosis and alveolar bone loss and tooth loss.

Vitamin D serum concentrations might affect periodontal disease both through an effect on bone mineral density (BMD) and through immunomodulatory effects. Vitamin D is well established as being essential for bone growth and preservation. A potential anti-inflammatory effect of vitamin D is supported by an increasing amount of literature. The active metabolite of 25-hydroxyvitamin D, 1,25dihydroxyvitamin D, has been found to inhibit cytokine production and cell proliferation.

Low serum levels of vitamin D have been linked with a loss of periodontal attachment. Data from over 11,000 subjects were analyzed for serum vitamin D levels and attachment loss. In subjects less than 50 years of age, there was no signiﬁcant association reported between vitamin D levels and attachment loss. In patients 50 years or older, serum vitamin D levels were inversely associated with attachment loss for men and women. It was concluded that the increased risk for periodontal disease might be attributable to low levels of vitamin D, which would reduce bone mineral density, or to an immunomodulatory eﬀect.

In van der Putten et al study, based on the literature available to date, the association of vitamin D, and calcium deﬁciencies with periodontal disease in elderly people is essentially still unknown and not well researched. To produce conclusive evidence on the subject of this systematic literature review, longitudinal cohort studies and follow-up randomized controlled trials are needed

The aim of this study is to explore chronic periodontitis status and serum vitamin D and calcium concentrations in Syrian males and compare these figures with matched healthy volunteers with no periodontitis.

ELIGIBILITY:
First group (Chronic Periodontitis) inclusion criteria:

1. Male patients
2. Patients are suffering from chronic periodontitis
3. Patients do no have systemic diseases
4. Patients should have 20 teeth at least
5. 30 year old at least

Second group (Healthy Volunteers) inclusion criteria:

1. Male individuals
2. With no systemic diseases or periodontitis
3. 30 year old at least
4. 20 teeth at least for each participant

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who are referred to the Periodontics Department at University of Damascus Dental School (Damascus, Syria) will be recruited in this research project. Healthy volunteers will be invited to participate in this research.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2014-05; Primary Completion 2015-08 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Serum Vitamin D concentration | One time assessment, within 24 hours before delivering any treatment
Serum Calcium concentration | One time assessment, within 24 hours before delivering any treatment

SECONDARY OUTCOMES:
Pocket Depth | One time assessment once sample recruitment has completed and within 24 hours before delivering any treatment.
Bleeding on Probing | One time assessment once sample recruitment has completed and within 24 hours before delivering any treatment.
Clinical Attachment Loss (CAL) | One time assessment once sample recruitment has completed and within 24 hours before delivering any treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Alharissi, DDS MSc, Principal Investigator — PhD student, Department of Periodontics, University of Damascus Dental School, Damascus; Suleiman Dayoub, DDS MSc PhD, Study Chair — Associate Professor of Periodontics, Department of Periodontics, University of Damascus Dental School, Damascus; Rowaida Saymeh, DDS MSc PhD, Study Director — Professor of Periodontics, Department of Periodontics, University of Damascus Dental School, Damascus
Locations (1):
- Department of Periodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Chapuy MC, Meunier PJ. [Calcium and vitamin D3, a prevention of femoral neck fractures in elderly women]. Presse Med. 1993 Apr 10;22(13):615-6. No abstract available. French. PMID 8390053
- [Background] Crowle AJ, Ross EJ, May MH. Inhibition by 1,25(OH)2-vitamin D3 of the multiplication of virulent tubercle bacilli in cultured human macrophages. Infect Immun. 1987 Dec;55(12):2945-50. doi: 10.1128/iai.55.12.2945-2950.1987. PMID 3119492
- [Background] Dennison DK, Van Dyke TE. The acute inflammatory response and the role of phagocytic cells in periodontal health and disease. Periodontol 2000. 1997 Jun;14:54-78. doi: 10.1111/j.1600-0757.1997.tb00192.x. No abstract available. PMID 9567966
- [Background] Jeffcoat M. The association between osteoporosis and oral bone loss. J Periodontol. 2005 Nov;76(11 Suppl):2125-32. doi: 10.1902/jop.2005.76.11-S.2125. PMID 16277585
- [Background] Kinane DF. Causation and pathogenesis of periodontal disease. Periodontol 2000. 2001;25:8-20. doi: 10.1034/j.1600-0757.2001.22250102.x. No abstract available. PMID 11155179
- [Background] Liu H, Komai-Koma M, Xu D, Liew FY. Toll-like receptor 2 signaling modulates the functions of CD4+ CD25+ regulatory T cells. Proc Natl Acad Sci U S A. 2006 May 2;103(18):7048-53. doi: 10.1073/pnas.0601554103. Epub 2006 Apr 21. PMID 16632602
- [Background] Ramanathan B, Davis EG, Ross CR, Blecha F. Cathelicidins: microbicidal activity, mechanisms of action, and roles in innate immunity. Microbes Infect. 2002 Mar;4(3):361-72. doi: 10.1016/s1286-4579(02)01549-6. PMID 11909747